CLINICAL TRIAL: NCT06956222
Title: The Effect of Hybrid Tele-rehabilitation Versus Standard Rehabilitation in Patients With Knee Osteoarthritis: A Single-blind Randomized Controlled Trial
Brief Title: The Effect of Hybrid Tele-rehabilitation Versus In Person Rehabilitation on Pain and Function in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Anfal Adnan Astek, Principle investigator, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tele-rehabilitation in OA
Record Dates: First submitted 2025-04-19; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Arm 1(hybrid tele-rehabilitation): Participants will receive in-person and video sessions of prescribed exercises.
  Arm 2 (standard rehabilitation): Participants will receive in-person sessions alone of prescribed exercises.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Tele-rehabilitation (Experimental): participants will receive one in-person and one video session per week for 8 weeks. Both sessions include the same exercise program delivered by a physiotherapist.
  Interventions: Other: Hybrid Tele-rehabilitation
- Standard Rehabilitation (Active Comparator): participants will receive two in-person sessions per week for 8 weeks. All sessions include an exercise program delivered by a physiotherapist.
  Interventions: Other: Standard Rehabilitation

INTERVENTIONS:
Other: Hybrid Tele-rehabilitation — In-person session: participants attend the session in physiotherapy clinic.They will receive exercises (attached in the study protocol document) under the physiotherapist's supervision, including watching and correcting exercise techniques.
  Video session: participants attend video session via Zoom platform (Zoom Video Communications, inc., USA), an accessible internet-based platform from any laptop or mobile device that offers a real-time video and audio communications. Participants will receive a Zoom link with a unique password. During the video session, the physiotherapist accesses from the clinic using a laptop, while participants are based at their home. Participants will receive exercises (attached in the study protocol document) with real time instructions from the physiotherapist. Instructions on downloading and accessing Zoom platform will be given to the participants in the first in-person session to ensure their readiness to access the Zoom platform.
  Arms: Hybrid Tele-rehabilitation
Other: Standard Rehabilitation — In-person session: participants attend the session in physiotherapy clinic.They will receive exercises (attached in the study protocol document) under physiotherapist's supervision, including watching and correcting exercise techniques.
  Arms: Standard Rehabilitation

SUMMARY:
People with knee osteoarthritis often need regular physiotherapy sessions to reduce pain and improve movement. Attendance of in-person sessions can be difficult because of travel and time. This study aims to learn if combining in-person and video sessions using Zoom works for people with knee osteoarthritis. The main questions it aims to answer are :

* Does combining in-person and video sessions improve pain and physical function in people with knee osteoarthritis?
* Does combining in-person and video sessions improve adherence to the exercise program?
* Are people satisfied with video sessions using Zoom?

The researchers will compare the use of one in-person session and one video session per week to the standard care of two in-person sessions per week.

Participants will :

* Attend either (one in-person and one video session per week) or (two in-person sessions per week) for 8 weeks.
* Perform exercise program that suits their needs during in-person and video sessions.
* Record the number of attended sessions over 8 weeks.
* Complete questionnaires about pain, physical function at the start and the end of the study.
* Complete questionnaire about usability and satisfaction at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate knee osteoarthritis.
* Age 40 to 80 years old.
* Body Mass Index < 34 kg/m2.
* Numeric pain rating scale > 4 out of 10.
* Pain for more than 3 months.
* Morning stiffness lasting < 30 minutes (standard clinical criteria of knee osteoarthritis)
* Pain and crepitus with active motion (e.g., walking, sit to stand, stair climbing) (standard clinical criteria of knee osteoarthritis)
* Access to the device with an internet connection.
* Ability to use electronic devices or smart phones.

Exclusion Criteria:

* Severe knee osteoarthritis and limited mobility or bonded to a wheelchair.
* Body Mass Index > 34 kg/m2
* On a waiting list for hip or knee surgery.
* Undergoing other forms of rehabilitation.
* Previous knee arthroplasty.
* Recent knee surgery within 6 months.
* Received cortisone injection within the previous 30 days.
* Rheumatoid arthritis, bilateral knee morning stiffness > 30 minutes.
* Unstable medical conditions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the pain intensity measured by Numeric pain rating scale | Baseline and after 8 weeks of the intervention
  The Numeric pain rating scale assesses the pain intensity using 11 points scale, where 0 indicates no pain and 10 indicates the worst pain
Change in physical function measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline and after 8 weeks of the intervention
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), a validated self reported questionnaire designed to assess the physical function of individuals with knee osteoarthritis. it consists of 17 items rated on a 5-points Likert scale ( 0=none, 4=extreme). Scores range from 0 to 68, in which higher scores indicate worse physical function
Changes in lower limb strength measured by 30 seconds chair stand test | Baseline and after 8 weeks of the intervention
  The 30 seconds chair stand test assesses the lower limb strength and functional performance. The participant will be asked to stand straight and return to sitting on a standard high chair as many times as possible within 30 seconds without using their arms. The total number of completed full stand will be recorded and a higher number indicates better lower limb strength and function.

SECONDARY OUTCOMES:
Exercise adherence measured by weekly adherence log | Weekly during 8 weeks of the intervention and at the end of the 8 weeks
  The weekly adherence log will be completed by the physical therapist to assess the participants adherence to either in person or zoom sessions. Adherence will be calculated as the number of calculated sessions over 8 weeks (2 sessions per week, 16 sessions). A higher number indicates better adherence to the exercise program.
Usability and satisfaction of Zoom based tele-rehabilitation measured by Tele-health Usability Questionnaire. | After 8 weeks of the intervention
  The Telehealth Usability Questionnaire (TUQ) is a validated patient-reported questionnaire to evaluate the usability of tele health services across six domains: usefulness, ease of use, interface quality, interaction quality, reliability, and satisfaction. It includes 21 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree). The higher scores indicate greater usability and satisfaction with Zoom tele-rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Anfal Astek, Principal Investigator — Department of Physical Therapy, Faculty of Medical Rehabilitation Sciences, King Abdulaziz University, Jeddah, Saudi Arabia
Locations (1):
- Department of Physical Therapy, Faculty of Medical Rehabilitation Sciences, King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared, including: Pain intensity scores (Numeric Pain Rating Scale), Functional scores (WOMAC function subscale, 30-Second Chair Stand Test), Exercise adherence log and Usability scores from the Telehealth Usability Questionnaire (TUQ)
Supporting Information: Study Protocol
Time Frame: Available after completion of the study and upon publication of the primary results
Access Criteria: Requests to access the de-identified data should be directed to the corresponding author

REFERENCES:
- [Background] Hinman RS, Kimp AJ, Campbell PK, Russell T, Foster NE, Kasza J, Harris A, Bennell KL. Technology versus tradition: a non-inferiority trial comparing video to face-to-face consultations with a physiotherapist for people with knee osteoarthritis. Protocol for the PEAK randomised controlled trial. BMC Musculoskelet Disord. 2020 Aug 7;21(1):522. doi: 10.1186/s12891-020-03523-8. PMID 32767989

DOCUMENTS (1):
  • Study Protocol (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT06956222/Prot_000.pdf